CLINICAL TRIAL: NCT02370342
Title: Robot-Assisted Laparoscopic HIFU (High-Intensity Focused Ultrasound) for Thermal Ablative Therapy of Small Renal Mass: Corroborating With Robot-Assisted Laparoscopic Partial Nephrectomy Specimens
Brief Title: Robot-Assisted Ultrasound for Thermal Ablative Therapy in Treating Patients With Small Kidney Masses Undergoing Surgery
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No funding
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4K-14-3; NCI-2014-02636 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 4K-14-3 (Other: USC Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2015-02-17; First posted 2015-02-24 (Estimated); Last update posted 2017-12-20 (Actual); Status verified 2017-12

CONDITIONS: Renal Carcinoma; Renal Mass
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — High-Intensity Focused Ultrasound Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Treatment (robot-assisted laparoscopic HIFU) (Experimental): Patients undergo robot-assisted laparoscopic HIFU thermal ablative therapy during partial nephrectomy.
  Interventions: Procedure: Robot-Assisted Laparoscopic Surgery; Procedure: High-Intensity Focused Ultrasound Ablation; Procedure: Therapeutic Laparoscopic Surgery; Device: Sonatherm 600i Ultrasonic Lesion Generating System

INTERVENTIONS:
Procedure: Robot-Assisted Laparoscopic Surgery — Undergo robot-assisted laparoscopic HIFU ablation
Procedure: High-Intensity Focused Ultrasound Ablation — Undergo robot-assisted laparoscopic HIFU ablation
  Other Names: HIFU
Procedure: Therapeutic Laparoscopic Surgery — Undergo laparoscopic partial nephrectomy
Device: Sonatherm 600i Ultrasonic Lesion Generating System — Device used for high-intensity focused ultrasound ablation
  Other Names: Sonatherm

SUMMARY:
This clinical trial studies a type of ultrasound called robot-assisted laparoscopic high-intensity focused ultrasound for performing thermal ablative therapy, or sound wave therapy, in treating patients with small kidney masses undergoing partial removal of the kidney. The robot-assisted ultrasound probe takes images of the kidney to help doctors locate the mass. The probe then uses high frequency sound waves to target and ablate (or destroy) the kidney mass, which may be a cancerous tumor or benign tissue. Surgery is then performed to remove the part of the kidney with the mass. Robot-assisted laparoscopic high-intensity focused ultrasound for thermal ablative therapy may be safer and help doctors see the tumor better when performing kidney surgery.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the efficacy of laparoscopic high-intensity focused ultrasound (HIFU) for the treatment of localized primary renal cancer to evaluate histological accuracy in successful ablation of the small renal mass, matched with intraoperative targeting.

SECONDARY OBJECTIVES:

I. To evaluate the safety and toxicity of laparoscopic HIFU for patients with primary renal cancer.

II. To evaluate the technical success of laparoscopic HIFU ablation.

OUTLINE:

Patients undergo robot-assisted laparoscopic HIFU thermal ablative therapy during partial nephrectomy.

After completion of study treatment, patients are followed up at 2 days, 2 weeks, 1 month, 6 months, 12 months, and then annually for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Presence of an enhancing solid renal mass =< 3.0 cm on radiological examination
* Tumors with a depth of not greater than 3.0 cm from a laparoscopically accessible surface-meaning no part of the tumor should be deeper than 3.0 cm from the surface
* Patients with solitary kidneys, bilateral renal tumors, compromised renal function (baseline creatinine > 1.4)
* Subjects must have given written informed consent
* Previous chemotherapy, and/or biological therapy for cancer are permitted provided that the acoustic properties of the tumor were not affected, but the subject should have recovered from the effects of these or of any prior surgery
* Subjects must be free of any clinically significant disease other than cancer that would interfere with the study evaluations
* Absolute neutrophil count (ANC) >= 1500 mm^-3
* Platelet count >= 100,000 mm^-3
* Hemoglobin >= 10 g/dl
* Prothrombin time (PT) =< 1.5 times upper limit of laboratory normal (ULN)
* Activated partial thromboplastin time =< 1.5 times ULN
* Urea and serum creatinine < 2.5 times ULN
* Total bilirubin < 1.5 times ULN
* Aspartate aminotransferase (AST) =< 3 times ULN
* Alkaline phosphatase < 2 times ULN, unless arising from bone

Exclusion Criteria:

* < 90% solid component on screening cross-sectional imaging
* Subjects deemed unsuitable candidates and not medically optimized for partial nephrectomy
* Tumors greater than 3.0 cm at their widest point
* Subjects with tumors lying < 1 cm from sensitive structures such as the ureter, renal vessels or adjacent bowel
* Subjects on concurrent anticoagulant, or immunosuppressive medication
* Subjects on anti-cancer medication whether biologic or pharmaceutical
* Women who are pregnant or nursing (pregnancy test to be performed within 24 hours prior to HIFU treatment)
* Subjects assessed by consultant anesthetist as unsuitable for general anesthetic
* Subjects having had prior ablation therapy on the same tumor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-12-18 (Estimated); Primary Completion 2018-12-18 (Estimated); Study Completion 2019-12-18 (Estimated)

PRIMARY OUTCOMES:
Planned ablation volume | Baseline (day of surgery)
  Ablation area of the kidney mass will be compared to the planned area under histopathologic review. Analyzed using a one-sided one sample T-test.
Necrosis volume | Baseline (day of surgery)
  Ablation area of the kidney mass will be compared to the planned area under histopathologic review. Analyzed using a one-sided one sample T-test.

SECONDARY OUTCOMES:
Tumor response | Up to 4 years
Disease free interval | From the date of treatment to the date of local or distant failure or until date of death, assessed up to 4 years
Time to local failure | From the date of treatment to the time to local failure, assessed up to 4 years
Time to distant failure | From the date of treatment to the time to documented metastatic disease, assessed up to 4 years
Overall success rate, measured as the combination of achieving local control of kidney cancer and demonstration of a favorable safety profile evidenced by enumeration of all adverse events by type, severity, and frequency | Up to 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Osamu Ukimura, Principal Investigator — University of Southern California
Locations (2):
- United States (2):
  - Keck Hospital of USC, Los Angeles, California
  - USC Norris Comprehensive Cancer Center, Los Angeles, California